CLINICAL TRIAL: NCT05928637
Title: An Open-label, Randomized, Multiple-dose, Three-way Crossover Study to Compare the Pharmacokinetic Characteristics and Safety Among D745, D759, and D150 in Healthy Subjects
Brief Title: A Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetics of D745, D759, and D150
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A125_03DDI2228
Record Dates: First submitted 2023-06-26; First posted 2023-07-03 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-06

CONDITIONS: Diabetes type2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): * Period 1: oral dose of D745 1 tablet.
  * Period 2: multiple oral dose of 1 tablet of D759 and 2 tablets of D150.
  * Period 3: multiple oral dose of 1 tablet of D745, 1 tablet of D759, and 2 tablets of D150.
  Interventions: Drug: D745, D759, D150
- Sequence 2 (Experimental): * Period 1: oral dose of D745 1 tablet.
  * Period 2: multiple oral dose of 1 tablet of D745, 1 tablet of D759, and 2 tablets of D150.
  * Period 3: multiple oral dose of 1 tablet of D759 and 2 tablets of D150.
  Interventions: Drug: D745, D759, D150
- Sequence 3 (Experimental): * Period 1: multiple oral dose of 1 tablet of D759 and 2 tablets of D150.
  * Period 2: oral dose of D745 1 tablet.
  * Period 3: multiple oral dose of 1 tablet of D745, 1 tablet of D759, and 2 tablets of D150.
  Interventions: Drug: D745, D759, D150
- Sequence 4 (Experimental): * Period 1: multiple oral dose of 1 tablet of D745, 1 tablet of D759, and 2 tablets of D150.
  * Period 2: multiple oral dose of 1 tablet of D759 and 2 tablets of D150.
  * Period 3: oral dose of D745 1 tablet.
  Interventions: Drug: D745, D759, D150
- Sequence 5 (Experimental): * Period 1: multiple oral dose of 1 tablet of D745, 1 tablet of D759, and 2 tablets of D150.
  * Period 2: oral dose of D745 1 tablet.
  * Period 3: multiple oral dose of 1 tablet of D759 and 2 tablets of D150.
  Interventions: Drug: D745, D759, D150
- Sequence 6 (Experimental): * Period 1: multiple oral dose of 1 tablet of D745, 1 tablet of D759, and 2 tablets of D150.
  * Period 2: multiple oral dose of 1 tablet of D759 and 2 tablets of D150.
  * Period 3: oral dose of D745 1 tablet.
  Interventions: Drug: D745, D759, D150

INTERVENTIONS:
Drug: D745, D759, D150 — QD, PO for 5 days

SUMMARY:
A clinical trial to compare the pharmacokinetic characteristics and safety among D745, D759, and D150 in healthy subjects

DETAILED DESCRIPTION:
An open-label, randomized, multiple-dose, three-way crossover study to compare the pharmacokinetic characteristics and safety among D745, D759, and D150 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult aged between 19 to 50 at screening
2. Weight ≥ 55kg(man) or 50kg(woman) with ideal body weight ±20%
3. Those who don't have clinically significant sign of diseases including history of 5 years.
4. Those who have been confirmed to be appropriate throughout screening health examination.
5. Those who voluntarily decide to participate in paper and agree to comply with the cautions after fully understand the detailed description of this clinical trial

Exclusion Criteria:

1. Those who have clinically significant disease or medical history of Hepatopathy, Renal dysfunction, Neurological disorder, Immunity disorder, Respiratory disorder, Genitourinary system disorder, Haemato-oncology disorder, Cardiovascular disorder or Psychical disorder.
2. Those who have a history of gastrointestinal surgery except simple appendectomy and hernia surgery which can interfere with drug absorption.
3. Those who have hypersensitivity to the main constituents or components of the investigational drug such as empagliflozin, metformin.
4. History of drug abuse.
5. Following results in clinical examination

   * Na < 135 mEq/L
   * K < 3.4 mEq/L
   * Ca > 10.5 mg/dL
   * AST or ALT > 1.25 times more than normal range
   * Total bilirubin > 1.5 times more than normal range
   * Total cholesterol > 1.5 times more than normal range
   * CKD-EPI < 60 mL/min/1.73 m2
   * HBsAg, HCV Ab, HIV Ag/Ab, Syphilis reagin test = positive
6. Under 5 min resting condition, systolic blood pressure ≥150 mmHg or or <90 mmHg, diastolic blood pressure ≥100 mmHg or <50 mmHg.
7. Those who have genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
8. Those who had medical examination requiring radioactive iodine contrast material injected through IV 48 hours prior to first IP administration.
9. Those who received investigational products or participated in bioequivalence test within 180 days before the first administration of clinical trial drugs
10. Those who donated whole blood within 60 days before the first date of administration and donated ingredients within 30 days or received blood transfusion in 30 days
11. Those who have used drugs that induce or inhibit drug metabolizing enzymes, such as barbiturates, or who have used drugs that may interfere with this study within 30 days before the first dosing day
12. Those who have used ETC, herbal medicinal preparations, OTC, vitamins 10 days before the first dosing date.
13. Those who exceed an alcohol, caffeine and cigarette consumption (caffeine> 5 cups/day, alcohol> 210g/week, smoking> 10 cigarettes/day) and not able to stop on smoking, caffeine and alcohol
14. Those who can't resist caffeine, drinking and smoking from 9am of administration day till discharge date.
15. Those who agree to contraception from the date of consent form was written till 2 weeks after the last dosing day and decide not to provide sperm during the participation of clinical trial
16. Woman who are pregnant or breastfeeding
17. Those who are deemed insufficient to participate in clinical study by investigators

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
AUCt | [0d, 12d, 24d] pre-dose, [2d, 14d, 26d] pre-dose, [3d, 15d, 27d] pre-dose, [4d, 16d, 28d] pre-dose, and 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12h, [5d, 17d, 29d] 24h
  Area under the concentration-time curve time zero to time
Cmax | [0d, 12d, 24d] pre-dose, [2d, 14d, 26d] pre-dose, [3d, 15d, 27d] pre-dose, [4d, 16d, 28d] pre-dose, and 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12h, [5d, 17d, 29d] 24h
  Maximum plasma concentration of the drug

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No